CLINICAL TRIAL: NCT05389111
Title: The Effect of Internal Discourses on the Perception of Trail-running Effort
Brief Title: Internal Discourses and Perception of Trail-running Effort
Acronym: UT4M2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 38RC22.0111
Record Dates: First submitted 2022-04-29; First posted 2022-05-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Physical Exertion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal discourses (Experimental): Introduction to internal discourses with a brief definition and key elements for implementation.
  Interventions: Other: Internal discourses
- Non-internal discourses (Sham Comparator): Introduction to the risks associated with the practice of activity in the mountain environment and practical tips to prevent the risks
  Interventions: Other: Non internal discourses

INTERVENTIONS:
Other: Internal discourses — This intervention will take place following the randomization performed at the V1 visit. It will be held in videoconference, will be led by a professional of the training field, specialist of the trail activity and trained in the use of mental strategies
  Arms: Internal discourses
Other: Non internal discourses — This intervention will take place following the randomization performed at the V1 visit. It will be held in videoconference, and will be conducted by a professional of the training field, specialist of the trail activity and coach of mountain guide
  Arms: Non-internal discourses

SUMMARY:
Determination of the effect of an intervention to develop the use of internal discourses on the perception of exercise during a sub-maximum effort following a trail running

DETAILED DESCRIPTION:
The practice of mountain running or "trail" is in full development in France and elsewhere in the world. This sport practice is associated with various constraints specific to the activity.

These constraints imposed on the body during the preparation, participation and recovery of this type of effort have an impact on multiple aspects of the individual (physiological, psychological, neurological...). Some studies have made it possible in each of the fields to advance the current knowledge about the trail-running environment. However, there are very few links between variables from different fields of research, even though these links are at the origin of the complex individual responses observed in the field.

Therefore it seems important to study the practice of trail running and its consequences on the individual, relying on a systemic approach of the individual who studies how psychological phenomena, physiological and cerebral interactions to predict behaviour and its health consequences.

The biopsychosocial models are based on this systemic approach and postulate that the perception of the individual's effort would be the main limit to the continuity of effort, performance because it causes the intensity to decrease - or even stop the effort - if this sensation becomes too strong.

Consequently, the study of certain interventions aimed at reducing this perception of effort, such as the one proposed in this project, seems to be an essential step to propose to the practitioners of this type of sport strategies allowing to practice in a healthy and efficient way.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-55 years
* Subjects available in Grenoble before and during the 15 days after the race
* Subjects subject to a social security scheme
* Subjects able to sign informed consent.
* Fluent in French

Exclusion Criteria:

* Cardiorespiratory, metabolic and neurological conditions
* People treated with anxiolytics and/or neuroleptics or ATCD for behavioural disorders
* Persons refusing to sign the participation consent
* Persons under guardianship
* Persons referred to in Articles L1121-5 to L1121-8 of the CSP

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Perception of effort during running. | 1 day
  Perception of Borg scale rated effort (0 no effort; 10, maximal effort) while running on a treadmill at sub-maximum intensity

SECONDARY OUTCOMES:
Psychological profiles of trail-running practitioners | 18 months
  Assessement of internal discourses use, pre-competitive anxiety, self-determined motivation to practice, achievement goals assessed by a questionnaire
Perception of effort depending on running distance | 18 months
  Comparison of the perception of effort (Borg scale rated effort (0 no effort; 10, maximal effort) while running) between subjects according to the distance of running
Link between the individual's physical level and perception of effort | 18 months
  Correlation between VO2max assessed during exercise testing in the laboratory and effort perception
Serological library | 18 months
  Comparison of circulating markers (e.g. BDNF, s100, creatine kinase, interleukins, to be defined a posteriori according to the physiological and cerebral effects observed) before and after the race
Performance on a cognitive task | 3 months
  Performance on a cognitive task performed on a computer
Brain activation during a cognitive task | 3 months
  Changes in brain oxygenation assessed by NIRS during a cognitive task
Perception of effort, attentional focus, self-efficacy and resources of self-control during a race situation | 1 day
  Change in perception of effort, attentional focus, self-efficacy and self-monitoring resources, assessed by a questionnaire during the race
Recovery kinetics of runners after a trail race. | 2 weeks
  Changes in the previous outcomes will be evaluated between the end of the race and 1-2 weeks after the race

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No